CLINICAL TRIAL: NCT06296979
Title: Effectiveness of Noninvasive Phrenic Nerve Neuromodulation in Subjects With Right Shoulder Pain and Hepatobiliary Visceral Comorbidity.
Brief Title: Effectiveness of Noninvasive Phrenic Nerve Neuromodulation in Shoulder Pain and Hepatobiliary Visceral Comorbidity.
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Seville (Other)
Responsible Party: Principal Investigator, Angel Oliva Pascual-Vaca, Doctor, University of Seville
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0881-N-23
Record Dates: First submitted 2024-02-23; First posted 2024-03-06 (Actual); Last update posted 2025-04-02 (Actual); Status verified 2025-03

CONDITIONS: Shoulder Pain
Keywords: phrenic nerve; Shoulder Pain; Nuromodulation
MeSH Terms: conditions — Shoulder Pain

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- USUAL PHYSIOTHERAPY (Active Comparator): the usual treatment of the center consisting of manual therapy, exercise and thermotherapy will be performed.
  Interventions: Procedure: common Physical therapy
- Transcutaneous electrical nerve stimulation (Experimental): The intervention group will receive the usual physiotherapy treatment at the health center and will also receive neuromodulation on the phrenic nerve at its exit through the anterior cervical region. The neuromodulation technique will be applied for 10 minutes.
  Interventions: Device: Phrenic nerve neuromodulation; Procedure: common Physical therapy

INTERVENTIONS:
Device: Phrenic nerve neuromodulation — The intervention group will receive the usual physiotherapy treatment at the health center and will also receive neuromodulation on the phrenic nerve at its exit through the anterior cervical region. The neuromodulation technique will be applied for 10 minutes.
  Arms: Transcutaneous electrical nerve stimulation
Procedure: common Physical therapy — the usual treatment of the center consisting of manual therapy, exercise and thermotherapy will be performed.

SUMMARY:
Pain, particularly shoulder pain, is a social and economic problem worldwide. Although visceral pathology is not yet taken into account in the diagnosis of these pains, it is likely that on numerous occasions the hepatobiliary visceral condition causes referred pain in the metameric area belonging to the shoulder due to the involvement of the phrenic nerve. Therefore, the aim of this project is to study the response of treatment by neuromodulation of the phrenic nerve for shoulder pain in patients with associated hepatobiliary pathologies, assessing the possible visceral involvement in the symptomatology.

DETAILED DESCRIPTION:
Approximately 80% of patients with liver disease suffer chronic pain and fatigue, which can lead to sensitization of the central and peripheral nervous system. Central sensitization is an increase in the responsiveness of neurons within the central nervous system, which can lead to generalized pain hypersensitivity. It has been shown that some lesions or inflammatory processes can trigger changes in the nervous system, generating persistent pain.

According to the theory of visceral referred pain, there are visceral and musculoskeletal stimuli that converge in higher centers capable of producing referred pain in regions where metameric innervation is shared. This raises the possibility that altered visceral mechanisms may provoke and chronify musculoskeletal pain.

According to this theory, people with structural or functional hepatobiliary pathologies may have referred pain in the right metameric territory of C2-C3-C4-C5, which may generate pain in the shoulder on the same side. This is due to the fact that the phrenic nerve sensitively innervates Glisson's capsule, so any affectation of this structure can generate afferent stimuli to the previously mentioned metameric levels.

The phrenic hypothesis plays a very important role today, having as its main "endorsement" the analgesic techniques of phrenic blockade used for shoulder pain after hepatectomy. In order to eliminate this post-operative shoulder pain, electrical or medical nerve blocks are used.

ELIGIBILITY:
Inclusion Criteria:

* Over 18 years of age.
* Subjects presenting right shoulder pain at the time of enrollment in the study.
* Presentation of a hepatobiliary visceral disorder that may justify the visceral etiology of the pain.
* That they agree to participate in the project by signing the informed consent form.

Exclusion Criteria:

* Patients with chronic pain due to other diseases such as malignant disease.
* Patients with rheumatic diseases.
* Cutaneous infection in the area of pain.
* Disease of neurological, traumatic, oncologic, or infectious origin that rules out the visceral origin of the pain.
* Uncooperative subject.
* Severe psychiatric disease.
* Loss of cognitive capacity.
* Contraindication to electrotherapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Estimated)
Dates: Start 2024-03-20 (Actual); Primary Completion 2026-12-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Numeric Pain Rating Scale | pre-treatment, 1 week, 4 week, 12 week.
  Perceived pain. Self-perceived pain intensity will be evaluated by a 0 to 10 Numeric Pain Rating Scale (NPRS), where 0 denotes no pain and 10 denotes the maximum possible pain.

SECONDARY OUTCOMES:
Algometry | pre-treatment, 1 week, 4 week, 12 week.
  Pain threshold to pressure at specific tender points of the shoulder: infraspinatus, deltoid and trapezius. PPT levels defined as the minimum pressure required to evoke pain will be assessed using a portable electronic pressure algometer. Change from baseline on algometry. The units of measurement of pressure pain will be Kg/cm2.
Goniometry passive | pre-treatment, 1 week, 4 week, 12 week.
  measurement of passive pain-free ranges of motion of flexion, internal rotation, external rotation and abduction of the right shoulder with a portable goniometer. the unit of measurement shall be the degree of movement.
Quick Dash questionnaire | pre-treatment, 1 week, 4 week, 12 week.
  Questionnaire that measures the function of the upper limb. It is composed of 11 items that are rated from 1 to 5, from least to most difficult to perform certain movements.
Goniometriy active | pre-treatment, 1 week, 4 week, 12 week.
  measurement of active pain-free ranges of motion of flexion, internal rotation, external rotation and abduction of the right shoulder with a portable goniometer. the unit of measurement shall be the degree of movement.

CONTACTS AND LOCATIONS:
Overall Officials: Ángel Oliva Pascual-Vaca, Dr, Principal Investigator — University of Seville
Locations (4):
- Spain (4):
  - Centro de Salud Ronda Histórica, Seville, Sevilla
  - Centro de Salud las Letanías, Seville, Sevilla
  - Centro de Salud Bellavista, Seville, sevilla
  - Centro de especialidades Morón de la Frontera, Morón de la Frontera, Seville

IPD SHARING:
Plan to Share IPD: No